CLINICAL TRIAL: NCT00557076
Title: Can Neural Adaptation After Severe Brain Injury be Facilitated?
Brief Title: The Efficacy of Familiar Voice Stimulation During Coma Recovery
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Shirley Ryan AbilityLab (Other); Northwestern Memorial Hospital (Other); Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B4951-R
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-03

CONDITIONS: Traumatic Brain Injury; Coma; Vegetative State; Minimally Conscious State
Keywords: Randomized Clinical Trial; Auditory Stimulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Coma; Persistent Vegetative State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Familiar Auditory Sensory Training (Experimental): FAST is a standardized passive auditory stimulation protocol. The patient is provided with customized recordings of stories told by people well known to the patient at least 1 year prior to injury. The stories represent specific events experienced by both the patient and the storyteller. The FAST protocol is provided on compact discs (CDs), using portable players and noise cancelling headphones, while patients were awake (ie, eyes open). Speakers were used for one patient not tolerating his headphones. The CDs were identical according to track duration, labeling, and administration procedures.
  Interventions: Behavioral: Familiar Auditory Sensory Training
- Sham Auditory Sensory Training (Sham Comparator): Placebo protocol is silence. Patients receive sham protocols for 10 minutes 4 times per day, with at least 2 hours in between, for 6 weeks.
  Interventions: Behavioral: Sham Auditory Sensory Training

INTERVENTIONS:
Behavioral: Familiar Auditory Sensory Training — Patient is provided with customized recordings of stories told by people well known to the patient at least 1 year prior to injury. The stories represent specific events experienced by both the patient and the storyteller. Patients received FAST for 10 minutes 4 times per day, with at least 2 hours in between, for 6 week.
  Arms: Familiar Auditory Sensory Training
Behavioral: Sham Auditory Sensory Training — The sham intervention is zero minutes of Familiar Auditory Sensory Training. Each day for 6 weeks 0 minutes of Familiar voice stimulation will be provided in 10 minute daily segments for 6 weeks. Each 10 minute recording is a digital recording of silence.
  Arms: Sham Auditory Sensory Training

SUMMARY:
The purpose of the study is to determine whether familiar vocal stimulation, provided during coma recovery, improves outcomes for persons who are unconscious after severe TBI. The primary hypothesis is that unconscious persons who receive standard rehabilitation (SR) plus a high-dose of Familiar Voice stimulation (FVs) compared to unconscious persons who receive SR plus a sham stimulation (Sham Group) will demonstrate:

1. Significantly more neurobehavioral functioning post-intervention compared to pre-intervention.
2. Using Functional Magnetic Resonance Imaging (fMRI), significantly higher average measures of volumetric activity in the whole brain, middle temporal gyrus bilaterally, primary auditory area, bilateral pre-frontal cortex, hippocampus and/or the cerebellum post-intervention compared to pre-intervention.

DETAILED DESCRIPTION:
Medical advances have improved the odds of surviving a severe traumatic brain injury (TBI) thereby increasing demands for rehabilitation. Medical rehabilitation management during coma recovery, however, has been hampered by a paucity of rigorous clinical trials examining rehabilitation effectiveness. This randomized clinical trial addresses this knowledge gap. The purpose of the study is to determine whether a high dose of familiar vocal stimulation (FVs) improves outcomes for persons who are unconscious after severe TBI. The research objectives are to:

1. Determine whether neural responses elicited with FVs improve neurobehavioral outcomes and/or elicit activations in expected regions.
2. Examine the relationship between neurobehavioral and neurophysiological responses to high doses of FVs during coma recovery.

There are two study cohorts and each group receives standard rehabilitation. The experimental group will be exposed daily to 40 minutes of FVs for 6 weeks. The Sham Group (Control Group 2) will receive 40 minutes of sham treatment, or silence, daily for 6 weeks.

The 40 minutes of FVs treatment will be provided in four 10 minute sessions. Each FV session will start with the subject hearing a familiar voice call the 'Subject's Own Name' aloud and then that same voice re-telling a memory or an event familiar to the subject. The person re-telling the event will be a person who experienced the event with the subject and who interacted with the subject on a daily basis for at least 1 year prior to injury.

ELIGIBILITY:
Inclusion Criteria:

* Severe brain injury of traumatic origin
* Non-brain penetrating gun shot wound
* Blunt trauma with subsequent closed head injuries such as diffuse axonal injury
* 18 years of age or older
* Unconscious for at least 28 days consecutively
* Medically Stable
* Does not have active seizures

Exclusion Criteria:

* History of brain injury
* More than 1 year post injury
* MRI is contraindicated (e.g., metal, titanium in brain)
* Ventilator dependent
* Cardiac contraindications
* The definition of traumatic brain injury excludes: (a) Lacerations or contusions of the face, eye, ear or scalp and fractures of facial bones with-out loss of consciousness; (b) Primary cause of injury is blunt trauma (e.g., contusion from blow to head) without subsequent closed head injuries such as contra coup or diffuse axonal injury; (c) Brain-penetrating gun shot wound; (d) Primary BI due to anoxic, inflammatory, infectious, toxic metabolic encephalopathies; (e) Cancer, brain infarction (ischemic stroke), intracranial hemorrhage (hemorrhagic stroke) aneurysms and arterio-venous malformations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa LB Pape, DrPH MA BS, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (3):
- United States (3):
  - The Rehabilitation Institute of Chicago, Chicago, Illinois
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia

REFERENCES:
- [Result] Pape TL, Rosenow JM, Harton B, Patil V, Guernon A, Parrish T, Froehlich K, Burress C, McNamee S, Herrold AA, Weiss B, Wang X. Preliminary framework for Familiar Auditory Sensory Training (FAST) provided during coma recovery. J Rehabil Res Dev. 2012;49(7):1137-52. doi: 10.1682/jrrd.2011.08.0154. PMID 23341285
- [Derived] Pape TL, Rosenow JM, Steiner M, Parrish T, Guernon A, Harton B, Patil V, Bhaumik DK, McNamee S, Walker M, Froehlich K, Burress C, Odle C, Wang X, Herrold AA, Zhao W, Reda D, Mallinson T, Conneely M, Nemeth AJ. Placebo-Controlled Trial of Familiar Auditory Sensory Training for Acute Severe Traumatic Brain Injury: A Preliminary Report. Neurorehabil Neural Repair. 2015 Jul;29(6):537-47. doi: 10.1177/1545968314554626. Epub 2015 Jan 22. PMID 25613986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a large urban community population and two acute rehabilitation hospitals. Community participants included patients not treated at the two acute rehabilitation hospitals. Acute rehabilitation programs included one U.S.
Pre-assignment Details: All patients with possible impairment in sound conduction were withdrawn prior to randomization. In total, 5 participants were withdrawn prior to randomization: 1 participant failed the auditory pathway screen, 2 participants recovered full consciousness, and 2 participants were placed in hospice by LAR. Therefore 16 participants were randomized.
Groups:
- FAST: high dose of familiar voice stimulation
  Familiar Voice Stimulation High Dose: The High Dose intervention is 1,680 minutes of Familiar Vocal Stimulation (FVs) provided in 40 minute daily segments at least 2 hours apart and for 6 weeks. Four CDs with 10 minutes of FVs preceded by the familiar voice calling out the subject's name, will be played (1 at a time) each day for 6 weeks providing 1,680 minutes of FVs.
- Sham: sham auditory stimulation
  Sham Auditory Stimulation: The sham intervention is zero minutes of Familiar Voice Stimulation. Each day for 6 weeks 0 minutes of Familiar voice stimulation will be provided in 10 minute daily segments for 6 weeks. Each 10 minute recording is a digital recording of silence.
Period: Overall Study
Arm/Group | FAST | Sham
Started | 8 | 8
Completed | 8 | 7 (One participant was withdrawn due to unblinding)
Not Completed | 0 | 1
Not completed — Unblinding | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FAST | Sham | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (11.0) | 34.4 (12.0) | 35.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Education Achieved at Injury [Number; unit: participants]
  High School Graduate or GED | 4 | 1 | 5
  Some College, No Degree | 1 | 3 | 4
  Bachelor Degree | 2 | 2 | 4
  Graduate or Professional Degree | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: DOCS Neurobehavioral Measure (DOCS = Disorders of Consciousness Scale) Change
Description: The primary outcome, the DOCS, is a reliable, valid and precise measure of global neurobehavioral functioning shown to remain stable over six weeks.The DOCS-25 starts with a systematic observation followed by administration of 25 sensory stimuli. Best responses to each stimulus are rated on a scale of 0 to 2 and total raw scores range from 0 (worst) to 50 (best). The DOCS change was calculated as the value at endpoint (6 weeks after Baseline) minus the value at Baseline.
Time Frame: Baseline and immediately after treatment ends (6 weeks after Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FAST: familiar voice stimulation
  FAST is a standardized passive auditory stimulation protocol described elsewhere.8 In brief, the patient is provided with customized recordings of stories told by people well known to the patient at least 1 year prior to injury. The stories represent specific events experienced by both the patient and the storyteller.
Arm/Group | FAST | Sham
Number analyzed (Participants) | 8 | 7
units on a scale | 13.5 (8.2) | 18.9 (15.6)
Statistical Analysis 1: Comparison: FAST vs Sham; The planned sample of 15 per group provided 80% power for a one-sided t-test to detect be-tween group endpoint differences in DOCS averages equivalent to an effect size of .91 (9 units). Clinically, this assumes that the FAST protocol would facilitate progression from one clinical state to another (e.g., vegetative (VS) to minimally conscious (MCS) states). The hypothesized effect was based on average DOCS change for a severe TBI sample receiving three weeks of acute rehabilitation; Test type: Non-Inferiority or Equivalence — Because 50% of the planned sample size was randomized, achieved power for the DOCS is 0.51; p = .465, t-test, 1 sided; DOCS scores were transformed to interval level measures using a many-faceted Rasch model anchored to values from a larger validation data set; Mean Difference (Final Values) = 5.4, 95% CI 2-sided [-11.1 to 21.9], Standard Error of Mean 7.00 — The mean difference between the baseline and endpoint DOCS test was compared between the FAST and Sham groups

2. Secondary Outcome: Coma Near Coma Scale
Description: The CNC scale measures arousal and awareness and test stimuli are administered to elicit a specified behavior. Presence/absence of this behavior is scored as 0, 2 or 4. Total raw scores range from 0 (consistently responsive) to 36 (extreme coma). The CNC change score was calculated as the 8th CNC measure minus the Baseline CNC measure. Since 2 CNC measurements were collected per week, the 8th CNC measure occurred in Week 4. To calculate the change, we used the eighth CNC measure because two patients (one per group) recovered full consciousness after the eighth CNC measure. In the second statistical analysis, all CNC measures were used to calculate the slope; this includes the Baseline CNC and CNC measures 2-8. Again, we used the first 8 CNC measures (instead of all 12 collected over 6 weeks of treatment) because two patients recovered full consciousness after the eighth CNC measure.
Time Frame: Baseline and after the 8th CNC assessment (4 weeks after Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAST | Sham
Number analyzed (Participants) | 8 | 7
units on a scale | 1.0 (0.6) | 0.25 (0.7)
Statistical Analysis 1: Comparison: FAST vs Sham; Power was not calculated for the CNC because the effect size was not published; Test type: Superiority or Other; p = 0.049, t-test, 1 sided; CNC scores were transformed to interval level measures using Rasch partial credit and Facets models. We then re-scaled these logits to 0-100 scales; Mean Difference (Final Values) = -.76, 95% CI 2-sided [-1.51 to -.00493], Standard Error of Mean .346 — The mean difference was calculated for each group using the eighth CNC measure minus the Baseline CNC measure
Statistical Analysis 2: Comparison: FAST vs Sham; Test type: Superiority or Other; p = .0022, t-test, 1 sided — To confirm that CNC results were not an anomaly at the final measurement and that the overall CNC response pattern was consistent, mixed-effect longitudinal models were conducted; Slope = -0.63, Standard Error of Mean 0.2 — The Baseline CNC measure and seven post-Baseline CNC measures (for a total of eight CNC measures) were used to calculate the slope

ADVERSE EVENTS:
Time Frame: Length of study participation, which was 6 weeks.
Description: A Data Safety Monitoring Plan was completed each day of study participation. Baseline vital signs/safety indicators were recorded on the Day 1 of admission. Changes in severity of vital signs/safety indicators were recorded. If changes were noted, the degree of severity was indicated by referring to the severity definition for each indicator.
Arm/Group | FAST | Sham
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
A limitation is achieved sample size. Given restrictive eligibility criteria, enrollment was lower than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes